CLINICAL TRIAL: NCT00151099
Title: Safety of Preoperative Oral Administration of a High Caloric Drink With Protein in Patients With Dysgnathia
Brief Title: Safety of Preoperative Oral Administration of a High Caloric Drink With Protein
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: There is no possibility to reach the target patient number within the set time frame
Sponsor: University Hospital Muenster (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 03-Anast-05
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2007-08

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: preoperative nutrition; postoperative nausea and vomiting; Dysgnathia; anesthesia
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Proteins

INTERVENTIONS:
Drug: high caloric drink with protein

SUMMARY:
The purpose of the study is to determine whether the oral administration of a high caloric drink with protein decreases the postoperative nausea and vomiting in patients with dysgnathia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with surgery for dysgnathia

Exclusion Criteria:

* Diabetes mellitus

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2005-09; Study Completion 2007-12 (Estimated)

PRIMARY OUTCOMES:
gastric residual at induction of anesthesia

SECONDARY OUTCOMES:
postoperative wellness
thermoregulation

CONTACTS AND LOCATIONS:
Overall Officials: Christiane Goeters, MD, Principal Investigator — Department of Anesthesiology and Intensive Care, University Hospital Muenster
Locations (1):
- Department of Anesthesiology and Intensive Care, University Hospital Münster, Münster, Germany